CLINICAL TRIAL: NCT02270775
Title: Traduction and Validation of the Central Sentitization Inventory Into French
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Other Study IDs: CSI-French
Record Dates: First submitted 2014-10-17; First posted 2014-10-21 (Estimated); Last update posted 2014-10-21 (Estimated); Status verified 2014-10

CONDITIONS: Fibromyalgia; Heathy Volunteers
Keywords: Questionnaire; Translation
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Time Perspective: Prospective

GROUPS / COHORTS (3):
- Fibromyalgia Patients: The central Sensitization questionnaire will be filled in by each patients included.
  After One week, patients will filled it the questionnaire again to study the reliability.
- Ankle sprain Patients: The central Sensitization questionnaire will be filled in by each patients included.
- Healthy Volunteers: The central Sensitization questionnaire will be filled in by each volunteer included.
  After One week, volunteers will filled it the questionnaire again to study the reliability.

SUMMARY:
The study will include a translation of the Central Sensisization Inventory into French and a cultural validation of the French version of the questionnaire (Reliability, discrimination and comparison with other questionnaires).

ELIGIBILITY:
Inclusion Criteria:

* Clinical Diagnosis of Fibromyalgia (Group 1)
* Clinical Diagnosis of a Acute of Subacute Ankle Spain (Group 2)
* Healthy Volunteer (Group 3)

Exclusion Criteria:

* Having any chronic pain (group 1 and group 2)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 3 groups:
  Fibromyalgia Patients (group 1) Acute or subacute Ankle Sprain (Group 2) Healthy Volunteers (Group 3)
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2014-10; Primary Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Reliability of the French version the Central Sensitization Inventory Score | 1 week

CONTACTS AND LOCATIONS:
Locations (1):
- Cliniques Universitaires Saint-Luc, Brussels, Brussels Capital, Belgium